CLINICAL TRIAL: NCT01472198
Title: A Phase 2 Randomized, Double-Blinded, Placebo-Controlled Study to Evaluate the Efficacy and Safety of GS-6624 Combined With Gemcitabine as First Line Treatment for Metastatic Pancreatic Adenocarcinoma
Brief Title: A Study to Evaluate the Efficacy and Safety of Simtuzumab Combined With Gemcitabine for Metastatic Pancreatic Adenocarcinoma
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Gilead Sciences (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: GS-US-324-0101
Record Dates: First submitted 2011-11-10; First posted 2011-11-16 (Estimated); Last update posted 2015-03-10 (Estimated); Status verified 2015-02

CONDITIONS: Pancreatic Cancer
Keywords: GSI; Gilead; Gilead Sciences; Pancreatic Cancer; PC; Gemcitabine; Phase 2; Phase II; GS-6624; Oncology; Monoclonal Antibody
MeSH Terms: conditions — Pancreatic Neoplasms; Neoplasms | interventions — simtuzumab; Gemcitabine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (4):
- Simtuzumab (open-label) (Experimental): Participants will receive simtuzumab 700 mg plus gemcitabine in cycles of 28 days for up to 3 years.
  Interventions: Drug: Simtuzumab; Drug: Gemcitabine
- Simtuzumab 200 mg (randomized) (Experimental): Participants will receive simtuzumab 200 mg plus gemcitabine in cycles of 28 days for up to 3 years.
  Interventions: Drug: Simtuzumab; Drug: Gemcitabine
- Simtuzumab 700 mg (randomized) (Experimental): Participants will receive simtuzumab 700 mg plus gemcitabine in cycles of 28 days for up to 3 years.
  Interventions: Drug: Simtuzumab; Drug: Gemcitabine
- Placebo (randomized) (Placebo Comparator): Participants will receive placebo to match simtuzumab plus gemcitabine in cycles of 28 days for up to 3 years.
  Interventions: Drug: Gemcitabine; Drug: Placebo to match simtuzumab

INTERVENTIONS:
Drug: Simtuzumab — Simtuzumab administered intravenously every 2 weeks for a total of 2 infusions (Days 1 and 15)
  Other Names: GS-6624
  Arms: Simtuzumab (open-label); Simtuzumab 200 mg (randomized); Simtuzumab 700 mg (randomized)
Drug: Gemcitabine — Gemcitabine 1000 mg/m^2 administered intravenously on Days 1, 8, and 15 of each 28-day cycle
  Other Names: Gemzar®
Drug: Placebo to match simtuzumab — Placebo to match simtuzumab administered intravenously every 2 weeks for a total of 2 infusions (Days 1 and 15)
  Arms: Placebo (randomized)

SUMMARY:
This study will compare the efficacy of simtuzumab (GS-6624) versus placebo in combination with gemcitabine in adults with pancreatic cancer. The treatment phase of this study will be comprised of 2 sequential parts: an open label treatment phase and a double-blinded treatment phase.

ELIGIBILITY:
Inclusion Criteria:

* Initial diagnosis of metastatic pancreatic cancer must have occurred ≤6 weeks prior to the completion of screening.
* The presence of measurable metastatic pancreatic cancer documented by contrast enhanced CT (or MRI) scan in addition to 1 of the following:

  1. Histological diagnosis of pancreatic adenocarcinoma confirmed by pathologist OR
  2. Pathologist confirmed histological/cytological diagnosis of adenocarcinoma consistent with pancreatic origin in conjunction with either:

     1. The presence of a mass in the pancreas OR
     2. A history of resected pancreatic carcinoma
* Measurable disease per RECIST (ver. 1.1)
* ECOG Performance Status of 0 or 1.
* Adequate hepatic, hematologic and renal functions.

Exclusion Criteria:

* A history or evidence of clinically significant disorder other than metastatic cancer of the pancreas.
* A diagnosis of pancreatic islet neoplasms.
* Subject has undergone major surgery other than diagnosis surgery within 4 weeks of randomization
* Presence of biliary obstruction requiring external drainage
* Brain metastases.
* Unstable cardiovascular function within the last 6 months of screening
* Clinically active liver disease, including active viral hepatitis (HBV or HCV) or cirrhosis
* Known HIV infection.
* Uncontrolled hypertension at Screening
* History or presence of any form of cancer, other than pancreatic cancer, within the 3 years prior to enrollment
* Prior or concurrent anti-tumor therapy (chemotherapy, antibody therapy, molecular targeted therapy, retinoid therapy, hormonal therapy) for the treatment of inoperable locally advanced or metastatic pancreatic cancer; prior radiotherapy and chemotherapy given as pre-operative neoadjuvant therapy or radio sensitizers for locally advanced pancreatic cancer are allowed.
* Uncontrolled systemic fungal, bacterial or viral infection
* Participation in an investigational drug or device trial with therapeutic intent within 30 days prior to study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 250 (Actual)
Dates: Start 2011-11; Primary Completion 2013-10 (Actual); Study Completion 2015-02 (Actual)

PRIMARY OUTCOMES:
Progression free survival | Up to 3 years
  Progression free survival is measured as time from date of randomization to the earliest event time of death regardless of cause or first indication of disease progression.

SECONDARY OUTCOMES:
Overall survival | Up to 3 years
  Overall survival is measured as time from date of randomization to death regardless of cause.
Objective response | Up to 3 years
  Objective response is assessed by the Response Evaluation Criteria In Solid Tumors (RECIST) criteria version 1.1 as complete response, partial response, stable disease, or progressive disease.

CONTACTS AND LOCATIONS:
Overall Officials: Zung Thai, MD, Study Director — Gilead Sciences
Locations (57):
- United States (44):
  - Birmingham Hematology and Oncology Associates, LLC, Birmingham, Alabama
  - University of South Alabama Mitchell Cancer Institute, Mobile, Alabama
  - Central Hematology Oncology Medical Group, Inc., Alhambra, California
  - Comprehensive Blood and Cancer Center, Bakersfield, California
  - California Cancer Associates for Research and Excellence (CCARE), Fresno, California
  - Pacific Shores Medical Group, Long Beach, California
  - UCLA Community Oncology Practice, Los Angeles, California
  - Stanford University Medical Center, Palo Alto, California
  - Wilshire Oncology Medical Group, Inc., Rancho Cucamonga, California
  - Sharp Health Care, San Diego, California
  - San Jose Medical Group, San Jose, California
  - Saint Mary's Regional Cancer Center, Grand Junction, Colorado
  - Hematology Oncology Associates, PC, Stamford, Connecticut
  - Florida Cancer Specialists, Tampa, Florida
  - Georgia Cancer Specialists, P.C., Atlanta, Georgia
  - Northwestern University, Chicago, Illinois
  - Oncology Hematology Care, Inc., Crestview Hills, Kentucky
  - Anne Arundel Medical Center, Annapolis Oncology Center, Annapolis, Maryland
  - West Michigan Cancer Center, Kalamazoo, Michigan
  - Providence Cancer Center Oncology and Hematology Care Clinic-Eastside Portland, Southfield, Michigan
  - Hematology and Oncology Associates at BridgePoint, Tupelo, Mississippi
  - Saint Joseph Oncology, Inc., Saint Joseph, Missouri
  - Washington University School of Medicine, St Louis, Missouri
  - Montana Cancer Institute Foundation c/o Montana Cancer Specialists, Missoula, Montana
  - Comprehensive Cancer Centers of Nevada, Henderson, Nevada
  - Saint Luke's-Roosevelt Hospital Center, New York, New York
  - Beth Israel Comprehensive Cancer Center, New York, New York
  - Duke University Medical Center, Comprehensive Cancer Center, Durham, North Carolina
  - Emerywood Hematology and Oncology, High Point, North Carolina
  - Oncology Hematology Care, Inc., Blue Ash, Ohio
  - PinnacleHealth, Harrisburg, Pennsylvania
  - Abington Hematology Oncology Associates, Inc., Willow Grove, Pennsylvania
  - Charleston Hematology Oncology Associates, PA, Charleston, South Carolina
  - South Carolina Oncology Associates, Columbia, South Carolina
  - Tennessee Cancer Specialists, Knoxville, Tennessee
  - Tennessee Oncology, PLLC, Nashville, Tennessee
  - Coastal Bend Cancer Center, Corpus Christi, Texas
  - University of Texas Southwestern Medical Center at Dallas, Dallas, Texas
  - San Antonio Military Medical Center, Fort Sam Houston, Texas
  - Center for Cancer and Blood Disorders, PC, Fort Worth, Texas
  - Joe Arrington Cancer Research and Treatment Center, Lubbock, Texas
  - Utah Cancer Specialists, Salt Lake City, Utah
  - Virginia Cancer Specialists, PC, Fairfax, Virginia
  - Virginia Cancer Institute, Richmond, Virginia
- Russia (13):
  - Republic Clinical Oncology Dispensary of the Ministry of Healthcare of Republic of Bashkortostan, Ufa, Bashkortostan Republic
  - Regional Oncology Dispensary, Ivanovo, Ivanovo Oblast
  - Medical Radiological Research Center of Russian Academy of Medical Sciences, Obninsk, Obninsk, Kaluga Oblast
  - Kursk Regional Oncologic Dispensary, Kursk, Kursk Oblast
  - Blokhin Cancer Research Center of Russia, Dept. of clinical pharmacology, Moscow, Moscow
  - State Institution "Blokhin Cancer Research Centre RAMS", Moscow, Moscow
  - Non-State Institution of healthcare "Central Clinical Hospital #1 OAO RZD, Moscow, Moscow
  - Non-state Healthcare Institution "N.A. Semashko Central Clinical Hospital #2 of JSC "Russian Railway, Moscow, Moscow
  - State Institution of Healthcare "Arkhangelsk Regional Clinical Oncology Dispensary", Arkhangelsk, Primorskiy (Maritime) Kray
  - Republican Clinical Oncologic Dispensary of Ministry of health of Republic Tatarstan, Kazan', Tatarstan Republic
  - State Budgetary Healthcare Institution "Nizhny Novgorod Regional Oncological Dispensary", Nizhny Novgorod
  - Budgetary Healthcare Institution of Omsk Region "Clinical Oncologic Dispensary", Omsk
  - Petrov Research Oncology Institute, Saint Petersburg

REFERENCES:
- [Derived] Benson AB 3rd, Wainberg ZA, Hecht JR, Vyushkov D, Dong H, Bendell J, Kudrik F. A Phase II Randomized, Double-Blind, Placebo-Controlled Study of Simtuzumab or Placebo in Combination with Gemcitabine for the First-Line Treatment of Pancreatic Adenocarcinoma. Oncologist. 2017 Mar;22(3):241-e15. doi: 10.1634/theoncologist.2017-0024. Epub 2017 Feb 28. PMID 28246206